CLINICAL TRIAL: NCT06824649
Title: SMART Use of Biologics in Chronic Rhinosinusitis With Nasal Polyposis
Brief Title: Biologics in Chronic Rhinosinusitis With Nasal Polyposis
Acronym: CRSwNP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00141846
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Chronic Sinusitis; Nasal Polyps
Keywords: Sinusitis; Biologics
MeSH Terms: conditions — Nasal Polyps; Sinusitis | interventions — Biological Factors

STUDY DESIGN:
Masking Description: The laboratory analyzing the samples will be blinded to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dupilumab (Active Comparator)
  Interventions: Biological: Biologic Agents
- Omalizumab (Active Comparator)
  Interventions: Biological: Biologic Agents
- Mepolizumab (Active Comparator)
  Interventions: Biological: Biologic Agents

INTERVENTIONS:
Biological: Biologic Agents — Evidence by way of phase III clinical trials has shown efficacy of dupilumab, omalizumab, and mepolizumab to placebo, leading to regulatory approval and widespread clinical use. However, data from these clinical trials does not show universal improvement and ideal control of disease across all patients with Chronic Sinusitis with Nasal Polyps (CRSwNP). Successful completion of this trial will help answer some of the most pressing clinical questions related to biologics and CRSwNP. Specifically, findings will inform whether any one biologic has superior outcomes to another and whether clinicians can identify patients at baseline who are most likely to improve on biologic therapy.

SUMMARY:
The prevalence of Chronic Sinusitis with Nasal Polyps (CRSwNP) in the United States is estimated at roughly 4%, which equates to over 13 million Americans. Until recently, the only medical treatment options available for patients with CRSwNP were corticosteroids, with surgery reserved for medical failure. The development of biologic medications over the last 5 years has revolutionized the treatment of CRSwNP. Three biologic medications have been FDA approved and available for the treatment of CRSwNP: dupilumab, omalizumab, and mepolizumab. However, data from the clinical trials for these drugs do not show universal improvement across all patients with CRSwNP. In fact, there is a wide range of outcomes for patients in these trials. The result is that clinicians have no way of knowing which specific biologic would be the best option for any given patient, nor do they know whether biomarkers can be used to predict response to biologics. It is hoped that findings from this study will inform whether any one biologic has superior outcomes to another and whether clinicians can identify patients at baseline who are most likely to improve on biologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmed diagnosis of chronic rhinosinusitis with nasal polyposis using ICAR-21 (International Consensus Statement 20215) criteria
* Bilateral nasal polyposis visible on sinonasal endoscopy
* Nasal polyp score > 5
* Baseline SNOT-22 total score > 30
* Patient elects biologic therapy for the management of CRSwNP
* Capable of receiving all 3 biologic therapy medications.
* Treatment with intranasal mometasone ≥200 μg. once daily (or equivalent of another intranasal corticosteroid) for 1-month prior to baseline visit.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* Endoscopic sinus surgery within 6-months preceding enrollment / randomization.
* Oral corticosteroid use within 30-days preceding enrollment / randomization.
* Serum IgE level outside the dosing range for omalizumab (i.e., <30 IU/ml. or a weight-based dose with insufficient data to determine dose as per FDA dosing chart)
* Comorbid atopic dermatitis, urticaria, or any other condition that would require a specific biologic per the standard of care.
* Currently pregnant or plan to become pregnant within the 6 months after enrollment / randomization.
* Any previous treatment with any of the 3 biologic medications.
* Comorbid cystic fibrosis, CVID, or ciliary dyskinesia.
* Comorbid systemic inflammatory disorders (e.g., GPA, EGPA, Sarcoidosis, SLE)
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks for participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Disease-Specific Quality of Life | 24 weeks
  The 22-item SinoNasal Outcome Test (SNOT-22; ©2006, Washington University, St. Louis, MO) will serve as the primary outcome of interest for all study aims/objectives. The SNOT-22 survey is a CRS-specific QOL instrument containing 22 questions (total summarized score range: 0-110) with high internal consistency and high test-retest reliability. The SNOT-22 utilizes Likert scales numbering from 0 ("No problem") to 5 "Problem as bad as it can be"). The SNOT-22 has been shown to discriminate between subjects with CRS and healthy controls, as well as identify significant differences after both medical and surgical treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Soler, MD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: No